CLINICAL TRIAL: NCT01175239
Title: Gene Therapy for SCID-X1 Using a Self-inactivating (SIN) Gammaretroviral Vector
Brief Title: Gene Therapy for X-linked Severe Combined Immunodeficiency (SCID-X1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06MI10
Record Dates: First submitted 2010-07-29; First posted 2010-08-04 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2016-10

CONDITIONS: X-linked Severe Combined Immunodeficiency
Keywords: X-linked severe combined immunodeficiency, gene therapy; Patients will be enrolled following diagnosis and referral to Great Ormond Street Immunology Service.
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases | interventions — propeptide convertase 5, rat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single infusion of autologous CD34+ cells (Experimental)
  Interventions: Genetic: Single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) gammaretroviral vector pSRS11.EFS.IL2RG.pre

INTERVENTIONS:
Genetic: Single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) gammaretroviral vector pSRS11.EFS.IL2RG.pre — Single infusion of autologous CD34+ cells transduced with the self-inactivating (SIN) gammaretroviral vector pSRS11.EFS.IL2RG.pre

SUMMARY:
X-linked severe combined immunodeficiency (SCID-X1) is an inherited disorder that results in failure of development of the immune system in boys. This trial aims to treat SCID-X1 patients using gene therapy to replace the defective gene.

ELIGIBILITY:
Inclusion Criteria:

1. No HLA identical (A,B,C,DR,DQ) family donor and no HLA identical unrelated donor available within 3 months of diagnosis or patients whose underlying clinical problems and prognosis would be significantly compromised by chemotherapy conditioning (including persisting pneumonitis, protracted diarrhoea requiring parental nutrition, ongoing visceral viral infection (herpes viruses, HSV,VZV,CMV, EBV or adenovirus), systemic BCG infection, virus-induced lymphoproliferation.
2. Diagnosis of classical SCID-X1 based on immunophenotype (absent, or reduced numbers of non-functional T lymphocytes) and confirmed by DNA sequencing
3. Parental/guardian voluntary consent
4. Boys between the ages of 0 and 16

Max Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Immunological reconstitution | 1-18 months post-infusion,then annually
  * Immunophenotyping: detection of naïve CD3+ T-cell numbers, CD4, CD8, TCRαβ, TCRγδ, CD16+CD56+ NK & gamma chain expression. TRECs may be enumerated as surrogate marker for new thymic emigrants post-gene therapy
  * Lymphocyte proliferation assays to test function of T cells
  * Representation of TCR families by flow cytometry (Vβ phenotyping), & CDR3 PCR spectratyping (Vβ spectratyping) to monitor physiological & potentially pathological clonal expansions
  * Restoration of antibody production (IgA, IgM, IgG) & serological responses to vaccinations & natural infections.

SECONDARY OUTCOMES:
Incidence of adverse reactions | from consent until 5 years post-infusion of gene-modified cells
  At each scheduled visit, adverse events that might have occurred since the previous visit or assessment will be elicited from the patient/parent/guardian.
  The investigators will maintain a record of all adverse events/occurrences in patients participating in the clinical trial. This record will be noted in the patient's medical notes.
  Adverse events that have a causal relationship to the IMP (ARs) and SAEs will be recorded on the AE reporting section of the CRF.
Molecular characterisation of gene transfer | until 5 years post-infusion of gene-modified cells
  Quantification of transgene copy numbers is determined on sorted cell populations by real-time PCR methodology. Detailed integration analysis may be used to investigate specific clonal expansions.
Normalisation of nutritional status, growth, and development | until 5 years post-infusion of gene-modified cells
  Normalisation of nutritional status, growth, and development will be assessed at each follow-up visit by the investigator through clinical examinations.

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Thornhill SI, Schambach A, Howe SJ, Ulaganathan M, Grassman E, Williams D, Schiedlmeier B, Sebire NJ, Gaspar HB, Kinnon C, Baum C, Thrasher AJ. Self-inactivating gammaretroviral vectors for gene therapy of X-linked severe combined immunodeficiency. Mol Ther. 2008 Mar;16(3):590-8. doi: 10.1038/sj.mt.6300393. Epub 2008 Jan 8. PMID 18180772
- [Background] Cavazzana-Calvo M, Hacein-Bey S, de Saint Basile G, Gross F, Yvon E, Nusbaum P, Selz F, Hue C, Certain S, Casanova JL, Bousso P, Deist FL, Fischer A. Gene therapy of human severe combined immunodeficiency (SCID)-X1 disease. Science. 2000 Apr 28;288(5466):669-72. doi: 10.1126/science.288.5466.669. PMID 10784449
- [Background] Hacein-Bey-Abina S, Le Deist F, Carlier F, Bouneaud C, Hue C, De Villartay JP, Thrasher AJ, Wulffraat N, Sorensen R, Dupuis-Girod S, Fischer A, Davies EG, Kuis W, Leiva L, Cavazzana-Calvo M. Sustained correction of X-linked severe combined immunodeficiency by ex vivo gene therapy. N Engl J Med. 2002 Apr 18;346(16):1185-93. doi: 10.1056/NEJMoa012616. PMID 11961146
- [Derived] Clarke EL, Connell AJ, Six E, Kadry NA, Abbas AA, Hwang Y, Everett JK, Hofstaedter CE, Marsh R, Armant M, Kelsen J, Notarangelo LD, Collman RG, Hacein-Bey-Abina S, Kohn DB, Cavazzana M, Fischer A, Williams DA, Pai SY, Bushman FD. T cell dynamics and response of the microbiota after gene therapy to treat X-linked severe combined immunodeficiency. Genome Med. 2018 Sep 28;10(1):70. doi: 10.1186/s13073-018-0580-z. PMID 30261899
- [Derived] Hacein-Bey-Abina S, Pai SY, Gaspar HB, Armant M, Berry CC, Blanche S, Bleesing J, Blondeau J, de Boer H, Buckland KF, Caccavelli L, Cros G, De Oliveira S, Fernandez KS, Guo D, Harris CE, Hopkins G, Lehmann LE, Lim A, London WB, van der Loo JC, Malani N, Male F, Malik P, Marinovic MA, McNicol AM, Moshous D, Neven B, Oleastro M, Picard C, Ritz J, Rivat C, Schambach A, Shaw KL, Sherman EA, Silberstein LE, Six E, Touzot F, Tsytsykova A, Xu-Bayford J, Baum C, Bushman FD, Fischer A, Kohn DB, Filipovich AH, Notarangelo LD, Cavazzana M, Williams DA, Thrasher AJ. A modified gamma-retrovirus vector for X-linked severe combined immunodeficiency. N Engl J Med. 2014 Oct 9;371(15):1407-17. doi: 10.1056/NEJMoa1404588. PMID 25295500